CLINICAL TRIAL: NCT03664219
Title: Evaluation of the Neurosensory Disturbances After Inferior Alveolar Nerve Lateralization With and Without Isolation of the Simultaneously Placed Implants Using Collagen Membrane
Brief Title: Neurosensory Disturbances After Inferior Alveolar Nerve Lateralization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ibrahim hassan bashier garoushi, Director, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14422016472019
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Intervention Model Description: Atrophied posterior mandible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isolation of IAN nerve with collagen membrane (Active Comparator)
  Interventions: Other: isolation of IAN from implant with collagen membrane
- without isolation of the IAN with collagen (Experimental)
  Interventions: Other: isolation of IAN from implant with collagen membrane

INTERVENTIONS:
Other: isolation of IAN from implant with collagen membrane — comparing between the neurosensory disturbances with and without isolation of the inferior alveolar nerve from implant

SUMMARY:
Evaluation of the neurosensory disturbances after inferior alveolar nerve lateralization with and without isolation of the simultaneously placed implants using collagen membrane And measuring the stability of implants after placement .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with with atrophied posterior mandibular ridge
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence pathological lesions
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Neurosensory disturbances - sensation regaining over time subjective ( a scale 1-10 ) and objective checking the area | Year
  Assessing the sensation regaining over time subjective ( a scale 1-10 ) and objective checking the area of sensation regaining

SECONDARY OUTCOMES:
Stability - Osstell device to assess the primary stability of placed dental implant | Year
  Osstell device to assess the primary stability of placed dental implant after nerve lateraliztion